CLINICAL TRIAL: NCT05467228
Title: Laryngeal Vibro-tactile Stimulation as a Non-invasive Symptomatic Treatment for Spasmodic Dysphonia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not get funded
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KIN-2022-30628
Record Dates: First submitted 2022-07-12; First posted 2022-07-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Adductor Spasmodic Dysphonia; Abductor Spastic Dysphonia; Laryngeal Dystonia
Keywords: Adductor Spasmodic Dysphonia; Abductor Spastic Dysphonia; Laryngeal Dystonia; Vibtro-tactile stimulation
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Low dose / continuous VTS (Experimental): Low dose refers to receiving VTS 5 times/week for 20 minutes each; non-task-specific, constant stimulation during non-speech
  Interventions: Device: vibro-tactile stimulation (VTS)
- Low dose / speech activated VTS (Experimental): Low dose refers to receiving VTS 5 times/week for 20 minutes each; VTS during connected speech
  Interventions: Device: vibro-tactile stimulation (VTS)
- High dose / continuous VTS (Experimental): High dose refers to receiving VTS 7 times/week for 20 minutes each; non-task-specific, constant stimulation during non-speech
  Interventions: Device: vibro-tactile stimulation (VTS)
- High dose / speech activated VTS (Experimental): High dose refers to receiving VTS 7 times/week for 20 minutes each; VTS during connected speech
  Interventions: Device: vibro-tactile stimulation (VTS)

INTERVENTIONS:
Device: vibro-tactile stimulation (VTS) — To apply vibro-tactile stimulation, participants will use a wearable device. It contains two vibratory motors (Precision MicrodrivesTM, Model 307 - 100) that are low-voltage (~1V), non-invasive and will be located approximately above the lateral portions of the thyroid cartilage. For this protocol, they vibrate at frequencies between 40 - 100 Hz (i.e., 100 times per second

SUMMARY:
The general aim of the research is to provide scientific evidence that vibro-tactile stimulation (VTS) represents a non-invasive form of neuromodulation that can induce measurable improvements in the speech of patients with laryngeal dystonia (LD) - also called spasmodic dysphonia (SD).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Confirmed diagnosis of adductor or abductor LD for a minimum of 6 months.

Exclusion Criteria:

* Regular intake of benzodiazepines
* Cognitive impairment: score < 27 on the Mini-mental State Examination (MMSE).
* Identify with a neurological or musculoskeletal impairment affecting speech motor function. These impairments may include a form of: Dyskinesia, Dystonia other than LD, Essential Tremor, Huntington's Disease, Multiple System Atrophy, Muscle Tension Dysphonia, Parkinsonism, Progressive Supranuclear Palsy, Spasticity, Intracranial Neoplasm (brain tumor), Spinal Neoplasm, Cerebrovascular Accident (Stroke), Mild Traumatic Brain Injury, Intracranial Hemorrhage, Multiple Sclerosis.
* Non-English speaker. We will not enroll people who cannot speak English, because the voice assessment procedures (Test sentences, CAPE_V clinical rating) have only been validated for English speakers at this point.
* Pregnant people. We will not enroll pregnant people as the device used in this study is investigational.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-08 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in perceived speech effort (PSE) | 24 months
  Speaker will assess effort themselves and assign an score (range: 0-10 with a score of '10' indicating most severe effort)
Change in smoothed cepstral peak prominence (CPPS) | 24 months
  CPPS provides a measure of the strength of the fundamental frequency within background aperiodicity (physical unit is dB)
Change in speech quality vector (SQV) (%) | 24 months
  A derived measure designed to understand if a participant's voice symptom improvement occurs across objective (CPPS) and subjective measures of speech (PSE). It is based on the relative change between two time points

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States